CLINICAL TRIAL: NCT06499311
Title: Effect of Foot Reflexology Versus Acupressure on Sleep Disturbance and Hot Flashes in Postmenopausal Women
Brief Title: Reflexology Versus Acupressure on Sleep Disturbance and Hot Flashes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmeen Samir Abdelazeem Ali, Physical Therapist Specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC/012/005081
Record Dates: First submitted 2024-07-03; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Postmenopausal Flushing; Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant will have one identification number that will be used to assign participants into two equal groups in number (n=27), sequentially numbered index cards will be secured in opaque envelopes. Another assistant for the researcher will open the sealed envelope and will allocated the participants according to their groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A; Foot Reflexology (Experimental): Foot reflexology for 15 minutes, 3 sessions per week for 6 weeks will applied at the medical border just above the heel, also at associated reflex points associated with the adrenal, hypothalamus, pituitary glands, heart and lung via manual pressure at reflexology zone.
  Interventions: Other: Foot Reflexology
- Group B; Acupressure (Experimental): Acupressure for 21 minutes, 3 sessions per week for 6 weeks will applied at four acupoints points (Shenmen point at wrist crease, Sanyinjiao point; at both feet, and Fengchi point; at hairline within occipital region on dorsal neck surface), bilaterally in addition to one in midline at the top of nose on centerline between eyebrows ends (Yintang point).
  Interventions: Other: Acupressure

INTERVENTIONS:
Other: Foot Reflexology — Foot Reflexology is an alternative medical practice involving the application of pressure to specific points on the feet. It has been reported as a non-invasive complementary therapy that was addressed as an effective technique that is reported to reduce premenstrual symptoms.
  Arms: Group A; Foot Reflexology
Other: Acupressure — Acupressure is a sort of massage therapy, was addressed as an effective technique that is reported to reduce premenstrual symptoms. Acupressure is a well-known form of Traditional Chinese Medicine that is a component of alternative treatments.
  Arms: Group B; Acupressure

SUMMARY:
World health Organization (WHO) estimates that by 2030, 1.2 billion women will be over 50 years old. With a prevalence of 70%, a hot flash is the most distressing symptoms associated with menopause. Postmenopausal associated sleep disturbances could affect those women social activities and one's daily positive functioning. Therefore, some patients and their providers seek alternative treatments such as relaxation techniques, acupressure, yoga, reﬂexology, regular exercise, balanced nutrition, herbal supplements, appropriate clothing, and frequent showers, have been shown to be effective in reducing symptoms associated with depression. So, this study will be the first one in this issue. Therefore, it will have valuable benefits in physical therapy field and scientific research.

DETAILED DESCRIPTION:
Fifty-four postmenopausal women suffering from moderate to severe hot flashes diagnosed with hot flashes questionnaire, and sleep disturbances diagnosed with Pittsburgh quality sleep index >5. Their age ranged from 45-55 years old with their body mass index ranged from 25 to 30 kilogram per meter square. Outcome measures were Pittsburgh sleep quality index and Hot flashes questionnaire, both were conducted at baseline and after the end of the study program. after recruiting study population, they will be divided into two equal groups randomly. Group A; will received foot reflexology (medical border just above the heel, reflex points associated with adrenal, hypothalamus, pituitary glands, heart and lung via manual pressure at reflexology zone), for 15 minutes, 3 sessions per week for 6 weeks. Group B; will received acupressure ((Shenmen point, Sanyinjiao point, Fengchi point; Yintang point), for 21 minutes, 3 sessions per week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 45 to 55 years old.
* Their body mass index ranged from 25 to 3 kilograms per meter square.
* Postmenopausal women suffering from moderate to sever hot flashes assessed by Hot Flashes Questionnaire.
* Postmenopausal women suffering from sleep disturbances more than five assessed by Pittsburgh sleep quality index.

Exclusion Criteria:

* Any emotional stress during at least 6 months.
* Any pharmacological medicines lead to sleep disturbances.
* Any mental disorders affect their sleep cycle.
* Taking hormone replacement therapy for the past six months.
* Using herbal medicine to improve menopausal symptoms severity.
* Circular job in particular night shifts.
* Sensorineural problems in their feet.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study targeting Postmenopausal women.
Enrollment: 54 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Pretreatment and immediately Posttreatment.
  A reliable, validated, self-reported questionnaire for assessing sleep quality. It is available of validated Arabic form that consists of seven components, namely, subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over a 1-month time interval. It held a good internal consistency, and convergent, also divergent validity.
  Each component scores are derived, each scored 'zero' means no difficulty, to 'three' means sever difficulty. component scores are summed to gain the whole score range 'zero to twenty-one' Higher scores indicates worse sleep quality.

SECONDARY OUTCOMES:
Hot Flashes Questionnaire | Pretreatment and immediately Posttreatment.
  A valid and reliable measure for severity of hot flashes. It is an appropriately sensitive tool to negative changes over time, with its cut-points and minimally important differences could prove a useful tool in targeting important issues regarding therapeutic interventions, and monitoring management progress and response using a 0 (do not interfere) to 10 (completely interfere) point scale. A total score is computed by summing items. Higher scores indicate higher interference due to hot flashes and thus, greater impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Walid M Zidan, PHD, Study Chair — Head and Professor of Obstetrics and Gynecology Department
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt